CLINICAL TRIAL: NCT02039063
Title: A Phase 1/2 Study of Repeated Intravenous E6011 Administration in Japanese Subjects With Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: E6011-J081-101; 142543 (Other: JapicCTI)
Record Dates: First submitted 2014-01-09; First posted 2014-01-17 (Estimated); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2019-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — quetmolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (4):
- 1 (Experimental): E6011 2 mg/kg
  Interventions: Drug: E6011 2 mg/kg
- 2 (Experimental): E6011 5 mg/kg
  Interventions: Drug: E6011 5 mg/kg
- 3 (Experimental): E6011 10 mg/kg
  Interventions: Drug: E6011 10 mg/kg
- 4 (Experimental): E6011 15 mg/kg
  Interventions: Drug: E6011 15 mg/kg

INTERVENTIONS:
Drug: E6011 2 mg/kg
  Arms: 1
Drug: E6011 5 mg/kg
  Arms: 2
Drug: E6011 10 mg/kg
  Arms: 3
Drug: E6011 15 mg/kg
  Arms: 4

SUMMARY:
This study is a multicenter, open-label, uncontrolled, multiple ascending dose (MAD) study to evaluate mainly the safety and tolerability of 12-week repeated intravenous administration of E6011. A total of 24 subjects will enroll into four cohorts. Six subjects per cohort will receive repeated intravenous administration of E6011.

DETAILED DESCRIPTION:
This study consists of Screening Phase, Observation Phase, Treatment Phase, Extension Phase, and Follow-up Phase. Screening assessments will be performed between 42 to 2 days before study drug administration. Observation Phase assessments will be performed a day before or on a day of the initial administration to confirm the eligibility of subjects. The eligible subjects will receive the repeated intravenous administration of E6011. E6011 will be dissolved in physiological saline (nearly 100 mL) for approximately 30-minute infusion. During the Treatment Phase, for the first and second cohorts, E6011 will be administered every 2 weeks up to Week 10, a total of 6 times (with a double dose at Week 0). For the third and fourth cohorts, E6011 will be administered at Weeks 0, 1 and 2, then every 2 weeks up to Week 10, a total of 7 times. Under no safety concerns, Crohn's Disease Activity (CDAI) is less than 150 or a decrease in CDAI from the Observation Phase is greater than 70 and a subject intends to continue administrations, the subject will receive a total of 20 subsequent biweekly administrations (40 weeks) at stable dose (Extension Phase). Subjects will be hospitalized for 24 hours after the initial and second administrations for postdose monitoring and will have out-patient monitoring until 12 weeks after the initial administration. If hospitalization is difficult after the second administration, the subjects can be held at the hospital for 6 hours and then allowed to go home after confirmation of the safety. Subjects who roll over onto the Extension Phase will have continued monitoring until 52 weeks after the initial administration. When the subjects complete (Week 12 or Week 52) or discontinue the study, they will undergo an on-site follow-up 28 days after the study completion or discontinuation and an off-site follow-up or telephone interview 70 days after the final administration. The investigator will conduct full assessments of subjects safety next day of the second administration (24 hours after the second administration) to confirm presence of absence of study-related manifestations which may affect the study drug administration of next cohort. When the sponsor is informed of investigator's judgment on the sixth subject in each cohort, the appropriateness of next cohort will be judged based on the safety data available including the judgment of individual investigator on the next day of the second administration.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Japanese patients aged 20 to 64 years old at the time of informed consent.
2. Diagnosed with Crohn's disease based on the diagnostic criteria for Crohn's disease of the Health and Labor Sciences Research Grants "Research on Measures against Intractable Diseases (Inflammatory Bowel Disease)" Group (2012).
3. Mild to moderate severity at Observation Phase (CDAI between 150 and 450, based on the above diagnosis criteria for Crohn's disease).
4. History of aminosalycylic acid (5-ASA), salazosulfapyridine, cortical steroid, immunomodulators, infliximab or adalimumab treatment with no apparent effect, or unable to continue the treatment due to AEs (except for infliximab and adalimumab).
5. Consent to use contraception (both the subject and the subject's partner), if the subject is a a man capable of reproduction or a woman of childbearing potential.
6. Has voluntarily consented, in writing, to participate in this study.
7. Has been thoroughly briefed on the conditions for participation in the study, and is willing and able to comply with the conditions.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Abscess or suspected abscess found at Screening or Observation Phase (not applicable to perianal abscess).
2. Diagnosed with gastrointestinal epithelia dysplasia at Screening or Observation Phase.
3. Suspected of colitis other than Crohn's disease at Screening or Observation Phase (such as pseudomembranous colitis).
4. Symptomatic obstruction at Screening or Observation Phase.
5. Underwent intestinal resection within 24 weeks before the start of the study treatment, or planning to undergo intestinal resection in the next 52 weeks.
6. Newly started with Seaton drainage within 12 weeks before Observation Phase.
7. Diagnosed with short bowel syndrome at Screening or Observation Phase.
8. Positive C.Difficile toxin test at Screening.
9. Prior history or current complication of malignant tumor, lymphoma, leukemia, or lymphoproliferative disease.
10. Immunodeficiency or history of HIV infection.
11. Infection requiring hospitalization or intravenous administration of antibiotics within 4 weeks before the start of the study treatment; or an infection requiring oral antibiotics within 2 weeks before the start of the study treatment.
12. History of tuberculosis or current complication of active tuberculosis.
13. History of serious allergy (shock, or anaphylactoid symptoms).
14. History of clinically important vascular edema, hematemesis, or hemoptysis.
15. History of acute myocardial infarction, cerebral infarction, cerebral hemorrhage, or arteriosclerosis obliterans.
16. History of clinically important vasculitis (such as mononeuritis multiplex).
17. In tests conducted at Screening, a positive finding for any of the following: human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B virus core antibody (HBc antibody), hepatitis B virus DNA (HBV DNA), hepatitis C virus antibody (HCV antibody), human T-lymphotrophic virus Type I antibody (HTLV-1 antibody), or syphilis screening. Except for the subject, if HBs antibody is only positive and is clear due to vaccination of Hepatitis B.
18. Any result other than negative in tuberculosis test (T-SPOT TB Test or QuantiFERON TB Gold Test) at Screening.
19. Findings indicating a history of tuberculosis on chest x-ray during screening.
20. Received a live vaccine within 12 weeks before starting the study treatment, or planning to receive a live vaccine before Week 52.
21. Planning to have surgery before Week 52.
22. Currently participating in another clinical trial, or used an investigational drug or investigational device, or participated in another clinical study, within 24 weeks of the start of the study treatment.
23. Judged to be ineligible to participate in this study by the investigator or sub-investigator

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04-05 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Japan (17):
  - Nagoya, Aichi-ken
  - Chikushino-shi, Fukuoka
  - Kurume, Fukuoka
  - Asahikawa, Hokkaido
  - Nishinomiya, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Morioka, Iwate
  - Sagamihara, Kanagawa
  - Tsu, Mie-ken
  - Urazoe, Okinawa
  - Takatsuki, Osaka
  - Minato-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Chiba
  - Fukuoka
  - Kyoto
  - Osaka

REFERENCES:
- [Result] Matsuoka K, Naganuma M, Hibi T, Tsubouchi H, Oketani K, Katsurabara T, Hojo S, Takenaka O, Kawano T, Imai T, Kanai T. Phase 1 study on the safety and efficacy of E6011, antifractalkine antibody, in patients with Crohn's disease. J Gastroenterol Hepatol. 2021 Aug;36(8):2180-2186. doi: 10.1111/jgh.15463. Epub 2021 Mar 31. PMID 33599356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 22 investigative sites in Japan from 05 April 2014 to 27 November 2017.
Pre-assignment Details: A total of 38 participants were screened, of which 10 were screen failures and 28 were enrolled to receive study treatment. As planned, combined data for Treatment Phase and Extension Phase is reported.
Groups:
- Cohort 1: E6011 2 mg/kg: Participants received E6011 2 milligram per kilogram (mg/kg), intravenous infusion for 30 minutes, every 2 weeks (double dose at Week 0) up to Week 10 in Treatment Phase. Participants who had no safety concerns, crohn's disease activity index (CDAI) was less than (<) 150 or clinical response (CR) greater than or equal to (>=) 70 and wished to continue with administrations had the opportunity to continue in the Extension Phase to receive 2 mg/kg, intravenous infusion for 30 minutes, every 2 weeks from Week 12 up to Week 52.
- Cohort 2: E6011 5 mg/kg: Participants received E6011 5 mg/kg, intravenous infusion for 30 minutes, every 2 weeks (double dose at Week 0) up to Week 10 in Treatment Phase. Participants who had no safety concerns, CDAI was <150 or CR >=70 and wished to continue with administrations had the opportunity to continue in the Extension Phase to receive 5 mg/kg, intravenous infusion for 30 minutes, every 2 weeks from Week 12 up to Week 52.
- Cohort 3: E6011 10 mg/kg: Participants received E6011 10 mg/kg, intravenous infusion for 30 minutes, at Week 0, 1, 2 and every 2 weeks up to Week 10 in Treatment Phase. Participants who had no safety concerns, CDAI was <150 or CR >=70 and wished to continue with administrations had the opportunity to continue in the Extension Phase to receive 10 mg/kg, intravenous infusion for 30 minutes, every 2 weeks from Week 12 up to Week 52.
- Cohort 4: E6011 15 mg/kg: Participants received E6011 15 mg/kg, intravenous infusion for 30 minutes, at Week 0, 1, 2 and every 2 weeks up to Week 10 in Treatment Phase. Participants who had no safety concerns, CDAI was <150 or CR >=70 and wished to continue with administrations had the opportunity to continue in the Extension Phase to receive 15 mg/kg, intravenous infusion for 30 minutes, every 2 weeks from Week 12 up to Week 52.
Period: Treatment Phase
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Started | 6 | 8 | 7 | 7
Completed | 3 | 6 | 5 | 5
Not Completed | 3 | 2 | 2 | 2
Not completed — Inadequate therapeutic effect | 3 | 2 | 1 | 1
Not completed — Progression of disease | 0 | 0 | 1 | 1
Period: Extension Phase
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Started | 1 (Only participants who met extension phase criteria started the period.) | 3 (Only participants who met extension phase criteria started the period.) | 5 (Only participants who met extension phase criteria started the period.) | 3 (Only participants who met extension phase criteria started the period.)
Completed | 1 | 2 | 2 | 2
Not Completed | 0 | 1 | 3 | 1
Not completed — Inadequate therapeutic effect | 0 | 1 | 2 | 0
Not completed — Progression of disease | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- Cohort 1: E6011 2 mg/kg: Participants received E6011 2 mg/kg, intravenous infusion for 30 minutes, every 2 weeks (double dose at Week 0) up to Week 10 in Treatment Phase. Participants who had no safety concerns, CDAI was <150 or CR >=70 and wished to continue with administrations had the opportunity to continue in the Extension Phase to receive 2 mg/kg, intravenous infusion for 30 minutes, every 2 weeks from Week 12 up to Week 52.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg | Total
Number analyzed (Participants) | 6 | 8 | 7 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (7.35) | 38.1 (12.33) | 39.9 (14.79) | 37.0 (8.16) | 36.8 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 3 | 7
  Male | 5 | 7 | 5 | 4 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6 | 8 | 7 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs was defined as adverse event (AEs) that emerged during the treatment, having been absent at pretreatment (Baseline) or re-emerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. An AE was defined as any untoward medical occurrence in a participants or clinical study participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. A SAE was defined as any untoward medical occurrence at any dose if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: Baseline up to Week 62 (70 days after last dose of study drug)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants
  TEAE | 6 | 6 | 7 | 3
  SAE | 1 | 1 | 5 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Change in Laboratory Parameters
Description: Clinical laboratory parameters included biochemistry, hematology, urinalysis and other screening test. Number of participants with clinically significant abnormalities in laboratory parameters which were deemed clinically significant by the investigator were reported.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change in Vital Sign Measurements
Description: Vital sign measurements included blood pressure (systolic and diastolic blood pressure) and pulse rate. Number of participants with clinically significant change in vital signs measurements which were deemed clinically significant by the investigator were reported.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-emergent Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: Number of participants with treatment-emergent clinically significant abnormal ECG findings which were deemed clinically significant by the investigator were reported.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Chest X-ray Findings
Description: Number of participants with abnormal chest X-ray findings were reported.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Neurological Findings
Description: Number of participants with neurological findings were reported.
Time Frame: Baseline up to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Mean Trough Serum Concentration of E6011 at Week 12 and 52
Time Frame: Week 12: Pre-dose; Week 52: Pre-dose
Population: The pharmacokinetic (PK) analysis set included participants who received at least 1 dose of study drug and had at least 1 serum E6011 concentration data. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here "n" was participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 3 | 6 | 5 | 5
microgram per milliliter (mcg/mL)
  Week 12 | 3.40 (3.74) | 26.1 (10.4) | 96.8 (60.3) | 146 (91.9)
  Week 52: number analyzed (Participants) | 1 | 2 | 2 | 2
  Week 52 | 10.8 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed. | 17.3 (2.90) | 105 (9.69) | 93.9 (46.8)

8. Secondary Outcome: Number of Participants With Serum Anti-E6011 Antibody at Week 12 and 52
Description: Number of participants with serum anti-E6011 antibody were reported.
Time Frame: At Week 12 and Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
Number analyzed (Participants) | 6 | 8 | 7 | 7
Participants
  Week 12 | 4 | 3 | 2 | 1
  Week 52 | 4 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 62 (70 days after last dose of study drug)
Description: As planned, combined safety data for E6011 administered in Treatment phase and Extension phase was reported.
Arm/Group | Cohort 1: E6011 2 mg/kg | Cohort 2: E6011 5 mg/kg | Cohort 3: E6011 10 mg/kg | Cohort 4: E6011 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/8 | 5/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/8 | 7/7 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: E6011 2 mg/kg (N=6) | Cohort 2: E6011 5 mg/kg (N=8) | Cohort 3: E6011 10 mg/kg (N=7) | Cohort 4: E6011 15 mg/kg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: E6011 2 mg/kg (N=6) | Cohort 2: E6011 5 mg/kg (N=8) | Cohort 3: E6011 10 mg/kg (N=7) | Cohort 4: E6011 15 mg/kg (N=7)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 2 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 2 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hyperaemia (Vascular disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No